CLINICAL TRIAL: NCT07258433
Title: A Randomized, Double-Blind, Placebo-Controlled, 6-Week Decentralised Trial Evaluating the Effects of PeptiSleep on Sleep Quality in Healthy Adults
Brief Title: Effects of PeptiSleep on Sleep Quality in Healthy Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nuritas Ltd (Industry)
Collaborators: Reputable Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: PEPSLE2
Record Dates: First submitted 2025-11-14; First posted 2025-12-02 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Sleep; Wearable Technology; Cortisol; Healthy Participants; Cognitive Abilities
Keywords: Sleep; Decentralised Study; Peptide Therapeutics; Protein Hydrolysates; Sleep Quality; Leeds Sleep Evaluation Questionnaire; Creyos; Oura; Wearable Technology
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Randomized, Decentralised, Double-Blind, Placebo-Controlled, Parallel-Design study conducted over 6-weeks
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PeptiSleep 250 mg/day (Experimental): One capsule to be consumed orally 30-60 minutes before bed
  Interventions: Dietary Supplement: PeptiSleep
- Microcrystalline Cellulose 250 mg/day (Placebo Comparator): One capsule to be consumed orally 30-60 minutes before bed
  Interventions: Dietary Supplement: Micro-crystalline cellulose

INTERVENTIONS:
Dietary Supplement: PeptiSleep — Rice Protein Hydrolysate
  Arms: PeptiSleep 250 mg/day
Dietary Supplement: Micro-crystalline cellulose — Placebo MCC micro-crystalline cellulose
  Arms: Microcrystalline Cellulose 250 mg/day

SUMMARY:
Examining the effects of PeptiSleep, a plant-based sleep aid, on sleep quality in healthy adults

DETAILED DESCRIPTION:
The primary aim of this is double-blind placebo-controlled parallel-design study is to measure the effects of PeptiSleep on sleep quality in healthy adults. PeptiSleep will be supplemented 30-60 minutes before bed as a single oral dose of 250mg for 6-weeks. A placebo group will also be included who will receive a matched dose of microcrystalline cellulose in identical capsules.

This trial incorporates a wearable sleep tracker to measure sleep biometrics which will be worn by participants for the duration of the study, as well as clinically validated questionnaires to measure sleep quality and a digital cognitive battery for to assess next day performance. The trial will be conducted over 6-weeks. 4 weeks of sleep tracking data will serve as a baseline prior to initiation of the supplementation period. The trial is fully decentralised.

The primary endpoint will measure the effects of PeptiSleep supplementation on responsive sleep quality via Leeds Sleep Evaluation Questionnaire versus a placebo from baseline to the end of the study period.

Secondary endpoints investigated during the trial will include changes in sleep biometrics (cardiac measures, sleep architecture, latency etc.) via Oura wearable, changes in comprehensive sleep quantity via Pittsburgh Sleep Quality Index (PSQI), next day readiness and next day performance via Creyos digital testing platform and safety and tolerability via adverse event reporting.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-65 at the time of enrollment.
* Generally healthy
* BMI 18.5 - 35.0kg/m2
* Willing and able to provide informed consent.
* Willing to consume one PeptiSleep or placebo capsule daily for 6 weeks.
* Willing to wear a sleep tracker continuously throughout the study period.
* Willing to complete all scheduled surveys and cognitive assessments on Days 0, 1, 2, and 3, at biweekly check-ins (Week 2 and Week 4), and at End-of-Study (Day 42).
* Willing to sync their wearable device data through the Reputable Health app and complete daily check-ins for compliance assessment
* Agree not to change current diet and/or exercise frequency or intensity during entire enrolment period.
* Agree to maintain a stable lifestyle and medication routines for at least 4 weeks prior to enrollment
* Agree not to use other medicines or supplements for sleep, stress, depression, or anxiety other than the test product during enrolment period.
* Agree to refrain from participation in another clinical trial during enrolment period.
* Agree to comply with Creyos digital platform data usage and privacy policy

Exclusion Criteria:

* Are currently pregnant, breastfeeding, or planning pregnancy during the study period.
* Are using prescription or over-the-counter sleep medications (e.g., zolpidem, melatonin >5 mg, benzodiazepines, CBD or antihistamines used for sleep, stress, depression, or anxiety within 4-weeks prior to enrolment.
* Have a current diagnosis of a chronic medical condition or illness (e.g., uncontrolled thyroid disease, diabetes, cardiovascular disease, major depressive disorder, or anxiety disorder requiring ongoing pharmacologic treatment) or a chronic sleep disorder, insomnia, restless leg syndrome, sleep apnoea.
* Are currently participating in any other clinical trial or who have participated in any other clinical trial during the past 4-weeks and any other sleep clinical trial during the past 3 months.
* Have a known allergy or sensitivity to any component of the investigational or placebo product
* Are shift workers or have highly irregular sleep/wake schedules that could confound study outcomes.
* Are unable or unwilling to comply with daily product use, wearable requirements, or survey/assessment completion.
* Have with significant non-wear time of their Oura device exceeding a 48- hour period
* Are using medications which induce CYP3A4 such as phenobarbital, phenytoin, rifampicin, St. John's Wort, and glucocorticoids.
* Are using prescription or OTC medications or supplements for sleep, stress, depression, or anxiety including CBD within one month prior to enrolment.
* Are using aromatherapy to help manage sleep, stress, depression, or anxiety within 4-weeks prior to enrolment.
* Are using a digital device (besides Oura) to help monitor or manage sleep during the study period.
* Have a current malignancy (excluding Basal Cell Carcinoma) or chemotherapy or radiotherapy treatment for malignancy within the previous 2 years.
* Have been diagnosed with or have consistent gastrointestinal issues that disrupt sleep.
* Have a history of renal function impairment
* Have with COPD or a chronic breathing disorder
* Are active smokers, nicotine use or drug (prescription or illegal substances) abuse.
* Have a chronic past and/or current alcohol use (>14 alcoholic drinks week)
* Are regularly taking stimulants (e.g., coffee, caffeine supplements, beverages containing caffeine) 5 hours before bed
* Are regularly consuming more than 500mg of caffeine per day
* Have any condition which in the opinion of the investigator makes the participant unsuitable for inclusion.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-12-29 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-03-28 (Estimated)

PRIMARY OUTCOMES:
Sleep Quality via Leeds Sleep Evaluation Questionnaire | Day 0 to Day 42
  Change from baseline to the end of the study period in Sleep Quality via Leeds Sleep Evaluation Questionnaire (LSEQ). The LSEQ comprises ten self-rating 100-mm-line analogue questions concerned with aspects of sleep and early morning behaviour. A visual analogue scale is used with two extreme states defined at the ends of the line (e. g. Tired = score of 0, Alert = score of 10). The subject responds by placing a vertical mark on the line to indicate his present self- evaluation.
  The four subscales are as follows:
  * The ease of getting to sleep (GTS), questions 1-3
  * The perceived quality of sleep (QOS), questions 4-5
  * The easy of awakening from sleep (AFS), questions 6-7
  * The integrity of behaviour following wakefulness (BFW), questions, 8-10

SECONDARY OUTCOMES:
Sleep Quality via Pittsburgh Sleep Quality Index | Day 0 to Day 42
  Change from baseline to the end of the study period in Sleep Quality via the Pittsburgh Sleep Quality Index (PSQI).
  The PSQI is a standardised self-rated questionnaire that assesses sleep quality and disturbances over a 1-month interval. It consists of 19 individual items, which generate seven component scores that reflect key aspects of sleep. Each component is scored on a scale from 0 to 3, where lower scores indicate no difficulty and higher scores indicate increasing difficulty. The seven component scores are summed to yield a global score ranging from 0 to 21, with higher global scores representing poorer overall sleep quality.
  The seven PSQI components are as follows:
  * Subjective Sleep Quality
  * Sleep Latency
  * Sleep Duration
  * Habitual Sleep Efficiency
  * Sleep Disturbances
  * Use of Sleeping Medication
  * Daytime Dysfunction
Heart Rate Variability via Wearable Technology | Day 0 to Day 42
  Change from baseline to the end of the study in heart Rate variability recorded as the time interval between two heartbeats in milliseconds between groups
Nocturnal Heart Rate via Wearable Technology | Day 0 to Day 42
  Change from baseline to the end of the study in the number of heart beats per minute while at rest and asleep between groups
Sleep Onset Latency via Wearable Technology | Day 0 to Day 42
  Change from baseline to the end of the study in sleep onset latency measured in minutes between groups
Sleep Architecture via Wearable Technology | Day 0 to Day 42
  Change from baseline to the end of the study in time spent in light, deep and REM phases of sleep between groups
Sleep Summary Metrics via Wearable Technology | Day 0 to Day 42
  Change from baseline to the end of the study in percentage Sleep score and Readiness scores between groups from 0-100 where 85 or higher is optimal, 70-84 is good and Under 70 is poor.
Safety and Tolerability via Adverse Event Reporting | Day 0 to Day 42
  Change from baseline to the end of the study period in safety and tolerability measured as the incidence ratio of adverse event reported between placebo and PeptiSleep
Feature Match Attention Test | Day 0 to Day 42
  Change from baseline to the end of the study period in attention between groups measured via feature match test on the Creyos cognitive digital platform. The test measured the number of correct matches within 90 seconds. Higher scores indicate better attention
Double Trouble Accuracy Test | Day 0 to Day 42
  Change from baseline to the end of the study period in accuracy and response time between groups via double trouble test on the Creyos cognitive digital platform. The test is scored by speed and accuracy in correctly identifying the colour of a word whilst ignoring the words meaning. Higher scored indicate better accuracy.
Token Search Memory Test | Day 0 to Day 42
  Change from baseline to the end of the study period in memory and cognitive performance between groups via token search Creyos cognitive digital test. The task score is determined by the maximum level completed and the users ability to solve a puzzle correctly without finding errors. Higher scores indicate better working memory and strategic ability
Visuospatial Reasoning via Number Ladder Test | Day 0 to Day 42
  Change from baseline to the end of the study period in visuospatial reasoning and cognitive performance between groups via the number ladder test on Creyos cognitive digital platform. The task score is based on the average number of boxes correctly remembered where higher scores indicate better visual memory.
Verbal Short Term Memory via Digit Span Test | Day 0 to Day 42
  Change from baseline to the end of the study period in verbal short term memory and cognitive performance between groups via digit span test on the Creyos cognitive digital platform. The score is calculated based on the longest sequence of digits correctly repeated, whereby higher scores indicate better verbal short term memory.

CONTACTS AND LOCATIONS:
Overall Officials: Mackenzie De Jesus, DHSc, MS, Principal Investigator — Reputable Health
Locations (1):
- Reputable Labs Inc., Wilmington, Delaware, United States

IPD SHARING:
Plan to Share IPD: No